CLINICAL TRIAL: NCT06771492
Title: Efficacy of Antibiotic Treatment for Patients With Chronic Low Back Pain and Modic Type I Changes - Randomized Placebo-controlled Trial
Acronym: ABBA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bart Koes (Other)
Collaborators: Erasmus University Rotterdam (Other)
Responsible Party: Sponsor-Investigator, Bart Koes, Prof. Dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-515824-35; 2024-515824-35-01 (EU CTIS Number)
Record Dates: First submitted 2024-11-21; First posted 2025-01-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: MSK Conditions; Chronic Low Back Pain (CLBP); Modic Changes
Keywords: Antibiotics; Amoxicillin; Low back pain (LBP); Modic changes; Randomized controlled trial
MeSH Terms: conditions — Low Back Pain | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic treatment (amoxicillin) (Experimental): A dose of 1000 mg (3 times a day) for a period of 100 days
  Interventions: Drug: Amoxicillin
- Placebo (Placebo Comparator): A dose of 1000 mg (3 times a day) for a period of 100 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Antibiotic treatment (amoxicillin) with a dosage of 1000 mg (3 times a day) for a period of 100 days
  Arms: Antibiotic treatment (amoxicillin)
Other: Placebo — Placebo with a dose of 1000 mg (3 times a day) for a period of 100 days
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if antibiotics (amoxicillin) work to treat chronic low back pain in adults. In some patients, this type of back pain may be caused by bacteria in the vertebrae, resulting in a condition known as "Modic type I change."

The main questions the trial aims to answer are:

* What is the efficacy (primary objective) of antibiotic treatment for patients with chronic low back pain and Modic type I changes?
* What is the cost-effectiveness (secondary objective) of antibiotic treatment for patients with chronic low back pain and Modic type I changes?

Researchers will compare amoxicillin to a placebo (a look-alike substance that contains no active drug) to see if amoxicillin works to treat chronic low back pain.

Participants in the trial will:

* Be invited for an MRI scan to determine if they have a Modic type I change; those who do will be included in the study.
* Take either amoxicillin or a placebo daily for 100 days.
* Take probiotics daily for 100 days to reduce the occurrence and impact of any side effects from the antibiotics.
* Attend clinic visits at baseline (the start), 4 weeks, 3 months, and 12 months for checkups and tests.
* Complete questionnaires at baseline, 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years.
* Chronic low back pain (i.e. duration >6 months) after a previous (MRI confirmed) disc herniation within the past 6 months to 2 years.
* At least 2 of the following questions should be answered with "Yes":

  * Does training and/or exercise increase your pain?
  * Is your sleep during the night disturbed due to your back pain?
  * Is it painful to turn over in bed at night?
  * Do you suffer from morning pain?
* The mean pain intensity should be at least 5 points on a 0-10 NRS-scale, calculated as the mean pain intensity of 3 indices: current pain, worst pain within the preceding two weeks, and the usual mean pain within the preceding two weeks.
* Modic Type I changes visible on the MRI-scan in the vertebrae adjacent to the previous herniated disc.

Exclusion Criteria:

* Received antibiotic treatment in the past month.
* Current pregnancy, lactation or pregnancy-wish.
* Severe physical or psychiatric co-morbidities.
* LBP resulting from a specific cause such as a tumor or fracture.
* Surgery or epidural injection in the past 6 months.
* Previous antibiotic course of 100 days.
* Contra-indication for amoxicillin use: allergy to penicillins/amoxicillin, cephalosporin or carbapenem; mononucleosis; leukemia; phenylketonuria (PKU)
* Contra-indication for MRI.
* Current use of any of the following medications: allopurinol, methotrexate, phenylbutazone or probenecid.
* Hepatic or renal (eGFR≤30) impairment.
* Inability to swallow capsules.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire (RMDQ) | The measurements are scheduled at baseline and at 3, 6 and 12 months follow-up.
  The primary outcome is pain and disability measured with the Roland Morris Disability Questionnaire (RMDQ). The scale ranges from 0-24 in which a higher score indicates higher disability. The RMDQ was also the primary outcome in the previous trials, and it is a recommended core outcome measure for trials in LBP.

SECONDARY OUTCOMES:
LBP-intensity (0-10 NRS-scale) | Measured at baseline, 3 months, 6 months and 12 months
  In the form of a questionnaire
Leg pain intensity (0-10 NRS-scale) | Measured at baseline, 3 months, 6 months and 12 months
  In the form of a questionnaire
Health-related quality of life (PROMIS-GH-10) | Measured at baseline, 3 months, 6 months and 12 months
  In the form of a questionnaire
Health-related quality of life (EQ-5D-5L) | Measured at baseline, 3 months, 6 months and 12 months
  In the form of a questionnaire
Self-reported number of days with sick leave | Measured at baseline, 3 months, 6 months and 12 months
  In the form of a questionnaire
Co-interventions (pharmacological and non-pharmacological) | Measured at baseline, 3 months and 12 months
  In the form of a questionnaire
Global perceived effect (7-point Likert scale) | Measured at 3 months, 6 months and 12 months
  In the form of a questionnaire
Patients' satisfaction with treatment (7-point Likert scale) | Measured at baseline, 3 months and 12 months
  In the form of a questionnaire
Success of blinding | Measured at 3 months and 12 months
  In the form of a questionnaire
Compliance | Measured at 3 months
  A pill count will be conducted
Pain self-efficacy (Pain Self-Efficacy Questionnaire) | Measured at baseline, 3 months, 6 months and 12 months
  In the form of a questionnaire
Sleep questionnaire (Pittsburgh Sleep Quality Index) | Measured at baseline, 3 months, 6 months and 12 months
  In the form of a questionnaire
Neuropathic pain (PainDETECT) | Measured at baseline, 3 months, 6 months and 12 months
  In the form of a questionnaire
Cost questionnaires (Medical Consumption Questionnaire) | Measured at 3 months, 6 months and 12 months
  In the form of a questionnaire
Cost questionnaires (Productivity Cost Questionnaire) | Measured at 3 months, 6 months and 12 months
  In the form of a questionnaire
Gut microbiome composition | Measured at baseline, 3 months, and 12 months
  The possible collateral impact of antibiotics on the microbiome would be investigated by comparing the abundance and diversity of microbial and resistome composition between patients in amoxicillin and placebo groups. They would be characterized using whole shotgun and functional metagenomic sequencing data (Dhariwal et al. Gut Microbes, 2023).
  In short, stools of the patients will be collected at baseline, 3 months, and 12 months. From these samples, the microbial DNA will be extracted using a commercial kit. Libraries for shotgun metagenomic sequencing would be prepared using Ilumina sequencing platform. Low quality and adapter sequences from paired-end reads will be filtered, and human DNA contaminant sequences will be discarded. The high-quality reads will be subjected to taxonomic classification. CARD antimicrobial resistance database will be used to annotate metagenomic reads.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Chiarotto A, Koes BW. Nonspecific Low Back Pain. N Engl J Med. 2022 May 5;386(18):1732-1740. doi: 10.1056/NEJMcp2032396. No abstract available. PMID 35507483
- [Background] Albert HB, Sorensen JS, Christensen BS, Manniche C. Antibiotic treatment in patients with chronic low back pain and vertebral bone edema (Modic type 1 changes): a double-blind randomized clinical controlled trial of efficacy. Eur Spine J. 2013 Apr;22(4):697-707. doi: 10.1007/s00586-013-2675-y. Epub 2013 Feb 13. PMID 23404353
- [Background] Braten LCH, Rolfsen MP, Espeland A, Wigemyr M, Assmus J, Froholdt A, Haugen AJ, Marchand GH, Kristoffersen PM, Lutro O, Randen S, Wilhelmsen M, Winsvold BS, Kadar TI, Holmgard TE, Vigeland MD, Vetti N, Nygaard OP, Lie BA, Hellum C, Anke A, Grotle M, Schistad EI, Skouen JS, Grovle L, Brox JI, Zwart JA, Storheim K; AIM study group. Efficacy of antibiotic treatment in patients with chronic low back pain and Modic changes (the AIM study): double blind, randomised, placebo controlled, multicentre trial. BMJ. 2019 Oct 16;367:l5654. doi: 10.1136/bmj.l5654. PMID 31619437
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CC, Chenot JF, van Tulder M, Koes BW. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. Eur Spine J. 2018 Nov;27(11):2791-2803. doi: 10.1007/s00586-018-5673-2. Epub 2018 Jul 3. PMID 29971708
- [Background] Agamennone V, Krul CAM, Rijkers G, Kort R. A practical guide for probiotics applied to the case of antibiotic-associated diarrhea in The Netherlands. BMC Gastroenterol. 2018 Aug 6;18(1):103. doi: 10.1186/s12876-018-0831-x. PMID 30078376
- [Background] Jafarnejad S, Shab-Bidar S, Speakman JR, Parastui K, Daneshi-Maskooni M, Djafarian K. Probiotics Reduce the Risk of Antibiotic-Associated Diarrhea in Adults (18-64 Years) but Not the Elderly (>65 Years): A Meta-Analysis. Nutr Clin Pract. 2016 Aug;31(4):502-13. doi: 10.1177/0884533616639399. Epub 2016 Apr 29. PMID 27130655